CLINICAL TRIAL: NCT00423930
Title: A Phase II Study of Radiotherapy (IMRT) + Cisplatin + Bevacizumab for Patients With Stage III/IV Head and Neck Cancers
Brief Title: Cisplatin, Bevacizumab, and Intensity-Modulated Radiation Therapy in Treating Patients With Stage III or Stage IV Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-130; MSKCC-06130; PFIZER-MSKCC-06130
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; tongue cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Bevacizumab; Cisplatin; Radiotherapy, Intensity-Modulated

ARMS (1):
- IMRT + cisplatin + bevacizumab (Experimental): This is a single-institution phase II study. The primary endpoint is to determine 2-year progression-free survival for patients with locally or regionally advanced HNSCC treated with concurrent intensity modulated radiation therapy (IMRT) + cisplatin + bevacizumab.
  Interventions: Biological: bevacizumab; Drug: cisplatin; Procedure: conventional surgery; Radiation: intensity-modulated radiation therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: cisplatin
Procedure: conventional surgery
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of head and neck cancer by blocking blood flow to the tumor. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving cisplatin and bevacizumab together with intensity-modulated radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving cisplatin and bevacizumab together with intensity-modulated radiation therapy works in treating patients with stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year progression-free survival of patients with stage III or IV squamous cell carcinoma of the head and neck treated with chemoradiotherapy comprising cisplatin, bevacizumab, and intensity-modulated radiotherapy.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Determine the median overall survival of patients treated with this regimen.

OUTLINE:

* Chemoradiotherapy: Patients receive cisplatin IV over 1 hour on days 1, 2, 22, 23, 43, and 44 and bevacizumab IV over 30-90 minutes on days 1, 22, and 43. Patients also undergo intensity-modulated radiotherapy on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47. Treatment continues in the absence of disease progression or unacceptable toxicity.

Between 3-4 months after completion of chemoradiotherapy, patients undergo evaluation. Patients with clinical evidence of residual, progressive, or persistent disease may be eligible to undergo neck surgery at the discretion of their physician.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Stage III/IV HNSCC without distant metastasis, previously untreated. Patients with stage II squamous cell carcinoma of the hypopharynx will also be eligible.
* Adequate renal function, with serum creatinine ≤ 1.5 mg/dL. Patients with serum creatinine > 1.5 mg/dL may be eligible if calculated creatinine clearance ≥ 55 ml/min by Cockcroft and Gault equation (or 24-hour urine collection).
* Age ≥ 18 years
* Karnofsky performance status ≥70%
* Adequate bone marrow function: absolute neutrophil count ≥ 1,500/μl, platelets ≥ 100,000/μl, hemoglobin ≥ 9 gm/dl
* Adequate hepatic function: Total bilirubin ≤ 1.5 X UNL (patients with Gilbert's syndrome as the cause of hyperbilirubinemia may be eligible if total bilirubin ≤ 2.5 X UNL), aspartate aminotransferase (AST) ≤ 2.5 X UNL, alanine aminotransferase (ALT) ≤ 2.5 X UNL, alkaline phosphatase ≤ 2.5 X UNL.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients must have ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy or radiation therapy for HNSCC
* Prior treatment with bevacizumab or other agents specifically targeting VEGF
* Other active malignancy, other than indolent malignancies which the investigator determines are unlikely to interfere with treatment or efficacy analysis. For example, patients with non-melanoma skin cancer, in situ carcinoma of the cervix, or prostate cancer within the no current biochemical (PSA) or radiologic evidence of disease may enroll.
* Patients with nasopharyngeal carcinoma
* Patients who will receive amifostine as part of the radiation treatment plan
* Patients with skin breakdown/ulceration (CTCAE version 3.0, grade 2 or higher).
* Patients with hearing loss requiring hearing aid or intervention (i.e. interfering in a clinical significant way with activities of daily living).
* Patients with multifocal peripheral sensory alterations or paresthesias (including tingling) interfering with function, per patient report (example: activities of daily living).
* History of arterial thromboembolic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, or myocardial infarction (MI) within the last 3 years.
* Urine protein: creatinine (UPC) ratio ≥ 1.0 at screening. A random urine sample is collected. Total protein (mg/dL) and spot creatinine (mg/dL) are ordered for this sample. The UPC ratio is calculated from the results of these tests.
* International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (aPTT) > 1.5 X upper limits of normal (UNL),
* Current use of warfarin, current use of heparin or low-molecular weight heparin, chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal antiinflammatory medications known to inhibit platelet function. Treatment with dipyramidole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and or cilostazol (Pletal) is not allowed.
* Patients with gross hemoptysis or hematemesis (defined as bright red blood of 1 teaspoon of more) within 1 month prior to Day 1 protocol treatment will be excluded from this trial. Patients with incidental blood mixed with phlegm are not excluded.
* Esophageal varices, non-healing ulcer, wound, or bone fracture are exclusion criteria. However, patients with skin breakdown overlying malignant neck lymphadenopathy may be eligible, at the discretion of the investigator.
* Anatomic lesion that increases the risk of serious hemorrhage, such as encasement or invasion of major blood vessels by primary tumor and/or by involved lymph nodes
* Blood pressure of > 150/100 mmHg
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* Clinically significant peripheral vascular disease
* History of bleeding diathesis or hemorrhagic disorder, or coagulopathy.
* Major surgical procedure or significant traumatic injury within 28 days prior to treatment with bevacizumab
* Core biopsy within 15 days prior to treatment with bevacizumab.
* Minor surgical procedures such as fine needle aspirations or placement of percutaneous gastrostomy tube (PEG) less than 7 days prior to treatment with bevacizumab
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior enrollment.
* Inability to comply with study and/or follow-up procedures
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G. Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- IMRT + Cisplatin + Bevacizumab: This is a single-institution phase II study. The primary endpoint is to determine 2-year progression-free survival for patients with locally or regionally advanced HNSCC treated with concurrent intensity modulated radiation therapy (IMRT) + cisplatin + bevacizumab.
  bevacizumab
  cisplatin
  conventional surgery
  intensity-modulated radiation therapy
Period: Overall Study
Arm/Group | IMRT + Cisplatin + Bevacizumab
Started | 44
Completed | 42
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Forty-four patients were enrolled on the study between November 20, 2006 and October 22, 2008. Two patients withdrew consent before receiving any treatment on the study.
Arm/Group | IMRT + Cisplatin + Bevacizumab
Number analyzed (Participants) | 44
Age, Continuous [Median (Full Range); unit: years] | 54 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 2 Years
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Percentage of Participants Experiencing Progression-free Survival at 2 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Bevacizumab
Number analyzed (Participants) | 42
percentage of participants | 75.9 [63.9 to 90.1]

2. Secondary Outcome: Overall Survival Rate: Percentage of Participants Who Survived
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMRT + Cisplatin + Bevacizumab
Number analyzed (Participants) | 42
percentage of participants | 88 [78.6 to 98.4]

ADVERSE EVENTS:
Arm/Group | IMRT + Cisplatin + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 11/42
Serious Adverse Events (participants affected / at risk) | 28/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Cisplatin + Bevacizumab (N=42)
ALT (Investigations) | 2
AST (Investigations) | 2
Alkaline Phosphatase (Investigations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Hyperbilirubinemia (Investigations) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine (Investigations) | 3
Death NOS (General disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophagitus (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 7
Fever (in the absence of neutropenia) (General disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hemoglobin/Anemia (Blood and lymphatic system disorders) | 7
Hemorrhage, Nose/Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemmorhage, Pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, Rectum (Gastrointestinal disorders) | 1
Hemorrhage, Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1
Hemorrhage/Bleeding, other (General disorders) | 3
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
INR (Investigations) | 1
Pneumonia (Infections and infestations) | 2
Leukoctyes (total WBC) (Investigations) | 6
Lymphopenia (Investigations) | 9
Mucositis - Oral Cavity (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 12
Neutrophils/Granulocytes (Investigations) | 8
Pain - Extremity/Limb (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain - other (General disorders) | 2
Pain - throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2
Peripheral arterial ischemia (Vascular disorders) | 1
Phosphate, low (Metabolism and nutrition disorders) | 2
Pleural effusion (non malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Prolonged QTc interval (Cardiac disorders) | 1
Pulmonary/upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Syncope (Nervous system disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 4
Urinary retention (Renal and urinary disorders) | 1
Valvular heart disease (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Weight loss (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IMRT + Cisplatin + Bevacizumab (N=42)
Fatigue (General disorders) | 42
Hyperglycemia (Metabolism and nutrition disorders) | 42
Anemia (Blood and lymphatic system disorders) | 42
Leukocytes (total WBC) (Investigations) | 42
Lymphopenia (Investigations) | 42
Mucositis - Oral Cavity (Gastrointestinal disorders) | 42
Pain - throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 42
Constipation (Gastrointestinal disorders) | 40
Nausea (Gastrointestinal disorders) | 40
Weight loss (Investigations) | 38
Hyponatremia (Metabolism and nutrition disorders) | 37
Hypoalbuminemia (Metabolism and nutrition disorders) | 36
Platelets (Investigations) | 33
Vomiting (Gastrointestinal disorders) | 32
ALT (Investigations) | 31
Neutrophils/granulocytes (Investigations) | 28
Tinnitus (Ear and labyrinth disorders) | 28
Diarrhea (Gastrointestinal disorders) | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Creatinine (Investigations) | 24
AST (Investigations) | 22
Hyperkalemia (Metabolism and nutrition disorders) | 18
Dermatitis Radiation (Injury, poisoning and procedural complications) | 17
Alkaline phosphatase (Investigations) | 16
Hypertension (Vascular disorders) | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 15
Mucosal infection (Infections and infestations) | 14
Oral Pain (Gastrointestinal disorders) | 14
Hypernatremia (Metabolism and nutrition disorders) | 14
Dehydration (Metabolism and nutrition disorders) | 12
Peripheral sensory neuropathy (Nervous system disorders) | 12
Fever (General disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 10
Blood bilirubin increased (Investigations) | 9
INR (Investigations) | 9
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 8
Trismus (Musculoskeletal and connective tissue disorders) | 8
Dry mouth (Gastrointestinal disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 7
Dysgeusia (Nervous system disorders) | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6
Urinary frequency/urgency (Renal and urinary disorders) | 6
Edema: limb (General disorders) | 5
Anxiety (Psychiatric disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 4
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 4
Cholesterol, high (Investigations) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Pain - middle ear (Ear and labyrinth disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 4
Confusion (Psychiatric disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
PTT (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Sinus bradycardia (Cardiac disorders) | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes